CLINICAL TRIAL: NCT05928039
Title: PATHFINDER: A Pragmatic, Active-comparator, Parallel-group, Randomized Trial to Evaluate the Optimal First-line Treatment Strategy for Moderate-to-Severely Active Ileal-dominant Crohn's Disease
Brief Title: PATHFINDER: Evaluating the Optimal First-Line Treatment Strategy for Moderate-to-Severely Active Ileal-dominant Crohn's Disease
Acronym: PATHFINDER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alimentiv Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB22-1641/RCT-01741
Record Dates: First submitted 2023-06-13; First posted 2023-07-03 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: This trial is a prospective, randomized, open-label, blinded-endpoint (PROBE) trial. The primary endpoint will be evaluated by a blinded, external central reviewer.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- TNFα antagonist (Active Comparator): Participants will receive either:
  * Infliximab 5 mg/kg intravenously [IV] at weeks 0, 2, 6, then 5 mg/kg every 8 weeks; OR
  * Adalimumab subcutaneously [SC] 160 mg at week 0, 80 mg at week 2, then 40 mg every 2 weeks
  Interventions: Biological: TNFa Antagonist - Infliximab; Biological: TNFa Antagonist - Adalimumab
- Anti-IL12/23 or anti-IL23 (Active Comparator): Participants will receive either:
  * Ustekinumab ~6 mg/kg IV x1, then 90 mg SC every 8 weeks; OR
  * Risankizumab 600 mg IV at weeks 0, 4, and 8, then 360 mg SC every 8 weeks
  Interventions: Biological: Anti-IL12/23 or anti-IL23 - Ustekinumab; Biological: Anti-IL12/23 or anti-IL23 - Risankizumab
- Anti-integrin (Active Comparator): Participants will receive either:
  * Vedolizumab 300 mg IV at weeks 0, 2, and 6, then every 8 weeks; OR
  * Vedolizumab 300 mg IV at weeks 0 and 2, then 108 mg SC every 2 weeks
  Interventions: Biological: Anti-integrin - Vedolizumab IV; Biological: Anti-integrin - Vedolizumab IV and SC

INTERVENTIONS:
Biological: TNFa Antagonist - Infliximab — • Infliximab 5 mg/kg intravenously [IV] at weeks 0, 2, 6, then 5 mg/kg every 8 weeks
  Arms: TNFα antagonist
Biological: TNFa Antagonist - Adalimumab — • Adalimumab subcutaneously [SC] 160 mg at week 0, 80 mg at week 2, then 40 mg every 2 weeks
  Arms: TNFα antagonist
Biological: Anti-IL12/23 or anti-IL23 - Ustekinumab — • Ustekinumab ~6 mg/kg IV x1, then 90 mg SC every 8 weeks
  Arms: Anti-IL12/23 or anti-IL23
Biological: Anti-IL12/23 or anti-IL23 - Risankizumab — • Risankizumab 600 mg IV at weeks 0, 4, and 8, then 360 mg SC every 8 weeks
  Arms: Anti-IL12/23 or anti-IL23
Biological: Anti-integrin - Vedolizumab IV — • Vedolizumab 300 mg IV at weeks 0, 2, and 6, then every 8 weeks
  Arms: Anti-integrin
Biological: Anti-integrin - Vedolizumab IV and SC — • Vedolizumab 300 mg IV at weeks 0 and 2, then 108 mg SC every 2 weeks
  Arms: Anti-integrin

SUMMARY:
There are currently three classes of biologic treatments approved in Canada for the management of moderate-to-severe Crohn's disease: anti-tumor necrosis factor [TNF] alpha, anti-integrin, and anti-interleukin [IL]-23 targeted agents. The purpose of this trial is to determine which of these three classes of biologics results in the highest percentage of patients with small bowel (ileal) Crohn's disease entering into endoscopic remission without needing corticosteroids at 1 year. Endoscopic remission means that the ulcers in the small bowel from Crohn's disease have healed. All treatments in this trial are approved by Health Canada. No experimental drugs will be included.

DETAILED DESCRIPTION:
This is a pragmatic, real-world trial of patients with moderate-to-severe, ileal-dominant Crohn's disease. At week 0, participants who meet the eligibility criteria will be randomized in a 1:1:1 ratio to a TNF antagonist; anti-integrin; or anti-IL23 targeted treatment. All interventions will be offered according to standard of care.

The dosing will be as follows:

TNFα antagonist

* Infliximab 5 mg/kg intravenously [IV] at weeks 0, 2, 6, then 5 mg/kg every 8 weeks; OR
* Adalimumab subcutaneously [SC] 160 mg at week 0, 80 mg at week 2, then 40 mg every 2 weeks

Anti-integrin

* Vedolizumab 300 mg IV at weeks 0, 2, and 6, then every 8 weeks; OR
* Vedolizumab 300 mg IV at weeks 0 and 2, then 108 mg SC every 2 weeks

Anti-IL23 targeted agents

* Ustekinumab ~6 mg/kg IV x1, then 90 mg SC every 8 weeks; OR
* Risankizumab 600 mg IV at weeks 0, 4, and 8, then 360 mg SC every 8 weeks

All treatments will be administered as part of the participant's routine care. All participants will be monitored per standard of care. Participants on corticosteroids at baseline will begin a steroid taper within 6 weeks of starting their biologic. At months 4, 8 and 12 participants will be evaluated for the Harvey Bradshaw Index (HBI), EuroQOL 5-domain questionnaire (EQ-5D), and be tested for C-reactive protein and fecal calprotectin concentrations. At month 12 patients will undergo a video-recorded ileocolonoscopy to determine if they have achieved endoscopic remission.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant, nonlactating females, 18 years of age or older. Females of childbearing potential must have a negative serum or urine pregnancy test prior to randomization
2. Established CD diagnosis by conventional criteria
3. Baseline colonoscopy within 3 months of the first day of the screening period, with photo or video documentation of at least one large ileal ulcer >5 mm and ileal segment SES-CD ≥4 (eligibility will be determined by local endoscopist, with subsequent confirmation by a CR at a later time, post enrolment)
4. HBI ≥5
5. Biologic-treatment naïve for CD-related therapies
6. Would otherwise have been eligible to start a biologic for moderate-to-severely active CD as part of their routine clinical care and for whom there is equipoise around which biologic class to start
7. Willing and able to participate fully in all aspects of this clinical trial, including adherence to study protocol and treatment algorithm
8. Written informed consent must be obtained and documented

Exclusion Criteria:

1. Condition(s) for which the biologics included in this study is contraindicated
2. CD-related complications such as symptomatic, endoscopically impassable strictures or abscesses that require imminent surgery (at investigator's discretion)
3. Participants with current or history of colonic dysplasia or neoplasia, toxic megacolon, or fulminant colitis
4. Recent bowel resection <3 months before screening
5. Active enteric infection (positive stool culture), including but not limited to bacterial (including C. difficile), viral, or parasitic enteric infections
6. Known active hepatitis B, hepatitis C, or human immunodeficiency virus infection
7. Active COVID-19 infection during the screening period
8. Tested positive as part of SOC for tuberculosis (TB) at screening by QuantiFERON® TB Gold Test, tuberculin skin test, or history of untreated latent or active TB
9. History of malignancy within 5 years of screening, except fully treated carcinoma in-situ of the cervix, fully treated and resolved nonmetastatic squamous or basal cell carcinoma of the skin
10. Active chronic or acute infections requiring treatment with systemic antibiotics, antivirals, antifungals, antiparasitics, or antiprotozoals during the screening period
11. Serious underlying disease other than CD that, in the opinion of the investigator, may interfere with the participant's ability to participate fully in the study
12. Not willing to withhold protocol-prohibited medications during the trial, or planned or anticipated use of any prohibited medications during screening
13. Received previously or currently receiving a TNF antagonist, anti-integrin, monoclonal antibody targeting IL-12/23 or IL-23, Janus kinase (JAK) inhibitors, or sphingosine 1 phosphate (S1P) receptor modulators (irrespective of indication)
14. History of alcohol or drug abuse that, in the opinion of the investigator, may interfere with the participant's ability to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Corticosteroid-free endoscopic remission | 1 year
  SES-CD ≤4, ileal segment SES-CD ≤2, and no ulcers in any segment >5 mm, off corticosteroids for ≥ 16 weeks

SECONDARY OUTCOMES:
CD-related complications | 1 year
  Composite of disease flare, obstruction, new fistula/abscess, CD-related hospitalization, CD-related surgery
Time to first Crohn's disease-related complication. | From date of randomization until the date of first documented Crohn's disease-related complication or date of death from any cause, whichever came first, assessed up to 12 months
  Composite of disease flare, obstruction, new fistula/abscess, CD-related hospitalization, CD-related surgery
Biomarker remission | Months 4, 8, and 12
  C-reactive protein (CRP) <5 mg/L and fecal calprotectin <250 µg/g, assessed in participants with elevated biomarkers at baseline
Corticosteroid-free clinical remission | Months 4, 8, and 12
  Harvey Bradshaw Index [HBI] ≤4 without exposure to systemic corticosteroids for ≥16 weeks prior to assessment
Treatment persistence | 1 year
  Duration of time from first biologic dose to discontinuation, the proportion of participants requiring a class switch, and the proportion of participants requiring dose optimization of biologic treatment or addition of rescue immunomodulators
Health-related quality of life after first-line biologic treatment | 1 year
  Quality of life at 1-year measured using EuroQol 5D (range 0 [worst imaginable health state] to 100 [best imaginable health state])
Safety of first-line biologic treatment | 1 year
  Unexpected AEs, severe AEs, drug and procedure-related AEs, any serious AEs (SAEs), any AEs leading to biologic discontinuation

CONTACTS AND LOCATIONS:
Locations (20):
- Canada (20):
  - University of Calgary, Calgary, Alberta
  - University of Alberta IBD Clinic, Edmonton, Alberta
  - GI Research Institute (G.I.R.I), Vancouver, British Columbia
  - West Coast Gastroenterology, Vancouver, British Columbia
  - Nova Scotia Health Victoria, Halifax, Nova Scotia
  - GNRR Digestive Clinics and Research Center Inc., Brampton, Ontario
  - Rajbir Rai Medical Corporation, Brantford, Ontario
  - McMaster University, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - West GTA Research Inc., Mississauga, Ontario
  - ABP Research Services Corp., Oakville, Ontario
  - Taunton Surgical Center, Oshawa, Ontario
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Thunder Bay Regional Health Research Institute, Thunder Bay, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - TIDHI Clinic, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Hôpital du Sacré-Cœur-de-Montréal, Montreal, Quebec
  - Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient information may be shared at the discretion the the trial steering committee and upon written request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available after completion of the trial and publication of results. Data will be retained for 15 years.

REFERENCES:
- [Derived] Hasskamp J, Meinhardt C, Timmer A. Anti-IL-12/23p40 antibodies for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2025 May 13;5(5):CD007572. doi: 10.1002/14651858.CD007572.pub4. PMID 40357993